CLINICAL TRIAL: NCT05505526
Title: Electroacupuncture for Women With Mixed Urinary Incontinence: a Sham-controlled Randomised Clinical Trial
Brief Title: Electroacupuncture vs Sham Electrocupuncture for Mixed Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shi Hangyu (Other)
Responsible Party: Sponsor-Investigator, Shi Hangyu, Principal Investigator, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Organization: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-174-KY
Record Dates: First submitted 2022-08-12; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Mixed Urinary Incontinence
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture (Experimental): Participants in EA group will receive treatment at bilateral Bladder Meridian (BL) 33 [Zhongliao], BL35 [Huiyang] and Spleen Meridian (SP) 6 [Sanyinjiao]. The EA treatment will last 30mins for each session, 3 sessions a week (ideally every other day) for a succession of 8 weeks.
  Interventions: Other: Electroacupuncture
- Sham electroacupuncture (Sham Comparator): Participants in SA group will receive treatment at bilateral sham BL33 [Zhongliao], sham BL35 [Huiyang] and sham SP6 [Sanyinjiao]. The SA treatment will last 30mins for each session, 3 sessions a week (ideally every other day) for a succession of 8 weeks.
  Interventions: Other: Sham electroacupuncture

INTERVENTIONS:
Other: Electroacupuncture — BL33 is located in the third posterior sacral foramen; BL35, 0.5 cun (≈10mm) lateral to the extremity of the coccyx; and SP6 posterior to the medial border of the tibia, 3 cun superior to the prominence of the medial malleolus. BL33 will be inserted by needles of 0.30×75mm size at the angle of 45°, inward and downward, till the depth of 60-70mm. BL35 will be inserted by needles of 0.30×75mm size, slightly outward and upward, till the depth of 60-70mm. SP6 will be inserted by needles of 0.30×40mm till the depth of 25-30mm. All the needles will be lifted, thrust and twisted evenly for three times, right after insertion, to induce the sensation of deqi. Electronic acupuncture apparatus (Yingdi KWD 808 I electro pulse acupuncture therapeutic apparatus, Changzhou Yingdi Electronic Medical Device Co., Ltd) will be connected to the three pairs of needles transversally, with continuous wave of 20 Hertz (Hz), electric current of 2-6.5 milliampere (mA) for BL33 and BL35, and 1mA-3.5mA for SP6.
  Other Names: EA
  Arms: Electroacupuncture
Other: Sham electroacupuncture — Sham BL33 is in the area of 1 cun (≈20mm) horizontally outside BL33; sham BL35, 1 cun (≈20mm) horizontally outside BL35; Sham SP6, in the middle of SP6 and tendons. The three pairs of acupoints will be inserted by needles of 0.30×40mm size to a depth of 2-3mm till the needles can stand still. No manipulations will be conducted, and the sensation of deqi will not be induced. Electronic acupuncture apparatus (Yingdi KWD 808 I electro pulse acupuncture therapeutic apparatus, Changzhou Yingdi Electronic Medical Device Co., Ltd) will be connected to the three pairs of needles transversally, with continuous wave of 20Hz and minimal electric current (ideally at a degree which participant can just percept). In about 30 seconds, the electric current will be turned down, leaving the indicator light and ticking sound on.
  Other Names: SA
  Arms: Sham electroacupuncture

SUMMARY:
The investigators plan to conduct this randomized sham-controlled clinical trial to evaluate the efficacy and safety of electroacupuncture (EA), compared with sham electroacupuncture (SA) on women with mixed urinary incontinence (MUI).

DETAILED DESCRIPTION:
MUI tends to present with more severe symptoms and put greater burden on the health of individual and economy of society. Current European Association of Urology (EAU) guideline on incontinence recommends to initiate treatment targeted at predominant component of MUI. Electroacupuncture has been proved not inferior to pelvic floor muscle training plus solifenacin in decreasing the 72-hour IEF and shows promise as an effective alternative for the treatment of MUI. The purpose of the study is to assess the efficacy and safety of electroacupuncture on mixed urinary incontinence among women.

ELIGIBILITY:
Inclusion Criteria:

* Female, 35 to 75 years old
* Diagnosed as mixed urinary incontinence
* Positive in cough stress test
* Experiencing persistent urinary incontinence for at least 3 months, and at least one episode for each of stress and urgent urinary incontinence in baseline screening
* Sign the informed consent form

Exclusion Criteria:

* Diagnosed as simple stress urinary incontinence, simple urgent urinary incontinence, overflowing urinary incontinence or neurogenic bladder, etc.
* Uncontrolled urinary tract infection with urinary pain and urge
* Urogenital system tumours and/or pelvic organ tumours
* Patients have taken drugs for urinary incontinence treatment or drugs possibly affect the function of lower urinary tract, or received non-drug treatment for urinary incontinence (i.e. electrical stimulation, bladder training, pelvic floor muscle training, and etc.) in the past one month
* History of surgeries for urinary incontinence and/or pelvic floor organs, including hysterectomy; Patients have pelvic organ prolapse ≥ II degree
* Residual urine ≥ 100ml
* Uncontrolled diabetes mellitus and severe hypertension
* Diseases affecting lower urinary tract function
* Severe heart, lung, brain, liver, kidney and hematopoietic system diseases, mental disorders and cognitive dysfunction
* Constrained or unable to complete movements like walking, going stairs up and down and running, etc.
* At pregnancy, breastfeeding or postpartum period for less than 12 months
* Cardiac pacemaker, metal allergy or strong fear of needle
* Patients have received acupuncture in the past 3 months

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2022-08-18 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the proportion of participants with at least 50 percent decrease from baseline in the mean 24-hour incontinence episodes. | week 8
  72-hour incontinence episodes dairy

SECONDARY OUTCOMES:
the proportion of participants with at least 50 percent decrease from baseline in the mean 24-hour incontinence episodes | week 4, 20, 32
  72-hour incontinence episodes dairy
the proportion of participants with at least 50 percent decrease from baseline in the mean 24-hour urgent incontinence episodes | week 4, 8, 20, 32
  72-hour incontinence episodes dairy
the proportion of participants with at least 50 percent decrease from baseline in the mean 24-hour stress incontinence episodes | week 4, 8, 20, 32
  72-hour incontinence episodes dairy
the change from baseline in the amount of urine leakage measured by the 1-hour pad test | baseline, week 8
  1-hour pad test
the change from baseline in the validated Chinese version of International Consultation on Incontinence Questionnaire-Short Form(ICIQ-SF) scores | week 4, 8, 20, 32
  data will be collected via International Consultation on Incontinence Questionnaire-Short Form(ICIQ-SF). The total score(0-21scores) is an accumulated scores from question 1 to 3. The higher the total score is, the severer the incontinence is.
the change from baseline in the validated Chinese version of the Overactive Bladder Questionnaire-Short Form scores | week 4, 8, 20, 32
  data will be collected via the Overactive Bladder Questionnaire-Short Form (0-15 scores). The higher the total score is, the severer the condition is.
incidence rate of any adverse events | up to 32 weeks
  adverse event will be documented as soon as it is reported during treatments and follow-ups
patients' expectation to treatment | baseline
  patients will be asked about their expected effect of the treatment via question: In your expectation, how is your incontinence like in a two month time. Five choices will be provided 1) much better; 2) slightly better; 3) I don't know; 4) no change; 5) worse.
blinding assessment | week 8
  patients will be asked whether they received electroacupuncture or sham electroacupuncture

CONTACTS AND LOCATIONS:
Overall Officials: Hangyu Shi, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Department of Acupuncture and Moxibustion, China Academy of Chinese Medical Sciences Guang'anmen Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No